CLINICAL TRIAL: NCT07087353
Title: A Randomized Controlled Trial Assessing the Efficacy of Remote Patient Monitoring in Patients Treated for a Moderate to Major Depressive Episode
Brief Title: Efficacy of Remote Monitoring in Patients Treated for Moderate to Major Depressive Episodes
Acronym: EC-102
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Resilience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-102; 2025-A01782-47 (Other: ANSM)
Record Dates: First submitted 2025-07-24; First posted 2025-07-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Mood Disorder (Depressive Episodes)
MeSH Terms: conditions — Mood Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Edra PRO
  Interventions: Device: Edra PRO
- Control (No Intervention): Standard care

INTERVENTIONS:
Device: Edra PRO — Remote monitoring software
  Arms: Intervention

SUMMARY:
Mood disorders like depression and bipolar disorder are widespread and cause serious psychological, cognitive, and social impairments, with a high burden on healthcare systems. Edra PRO is a digital medical device developed to support clinical decision-making and remotely monitor symptoms in psychiatric patients. The EC-102 randomized controlled trial will evaluate its impact compared to usual care on symptoms, quality of life, healthcare costs, comorbidities, and user adherence and satisfaction.

DETAILED DESCRIPTION:
Mood disorders such as depression and bipolar disorder affect a large portion of the global population and cause significant psychological, cognitive, and functional impairments, along with high healthcare costs. Despite available treatments, sustained remission is hard to achieve, and many patients experience persistent symptoms and treatment side effects. Continuous remote monitoring could improve care and outcomes. Edra PRO is a digital medical device designed for remote symptom tracking and clinical decision support in psychiatry. The EC-102 randomized controlled trial will assess the impact of Edra PRO versus usual care on symptoms, quality of life, healthcare costs, comorbidities, and user satisfaction and adherence.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old) meeting ICD-11 criteria for a moderate to severe major depressive episode
* Access to a personal smartphone and an internet connection, and cognitively able to use it independently

Exclusion Criteria:

* Pregnant women
* Individuals under legal guardianship or conservatorship
* Ongoing alcohol or drug abuse considered likely to interfere with study participation, as judged by the investigator
* Psychiatric or physical comorbidities (e.g., severe neurological or cardiovascular conditions) considered likely to interfere with participation or study results, at the discretion of the Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Response rate over a 6-month period. | Month 6
  Difference in response rates (%) between the intervention group and the control group

SECONDARY OUTCOMES:
Safety and absence of defects in Edra PRO over a 6-month period | Month 6
  Analysis of adverse events in both arms and reported device deficiencies in the intervention group
Impact of Edra PRO versus usual care on patients' quality of life | Month 6
  Short Form-36 questionnaire. Ranges from 0 to 100, with higher scores indicating better health-related quality of life.
Medico-economics impact of Edra PRO versus usual care | Month 6
  Analysis of cost of care

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Yrondi, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (6):
- France (6):
  - CHU Besançon, Besançon
  - CHU Grenoble Alpes, Grenoble
  - EPSM de VEndée, La Roche-sur-Yon
  - CHU de Lille, Lille
  - Cabinet Corinne MARIE, Lisieux
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No